CLINICAL TRIAL: NCT00115531
Title: Comparisons of the Reactogenicity and Immunogenicity in Ambulatory Elderly Subjects of a Standard-Dose Fluzone® (15 µg HA/Virus Strain) and a High-Dose (60 µg HA/Virus Strain) of a Trivalent Inactivated Influenza Virus Vaccine
Brief Title: Eldery High Dose TIV 2005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-100
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2007-02

CONDITIONS: Influenza
Keywords: Elderly, influenza, vaccine, parent protocol
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Arm 1 (Experimental): Standard Dose Influenza Vaccine Fluzone® (15 µg HA / viral strain; 45 µg/0.5 mL dose) will be administered to Arm 1: 200 subjects intramuscularly on day 0.
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Arm 2 (Experimental): High Dose Influenza Fluzone® Vaccine (60 µg HA / viral strain; 180 µg/0.5 mL dose) will be administered to Arm 2: 200 subjects intramuscularly on Day 0.
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Standard Dose Influenza Vaccine Fluzone® (15 µg HA / viral strain; 45 µg/0.5 mL dose) will be administered to Arm 1: 200 subjects intramuscularly on day 0.
  Arms: Arm 1
Biological: Trivalent inactivated influenza vaccine — High Dose Influenza Fluzone® Vaccine (60 µg HA / viral strain; 180 µg/0.5 mL dose) will be administered to Arm 2: 200 subjects intramuscularly on Day 0.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to compare a new higher-dose influenza virus vaccine to the standard dose vaccine in elderly adults who can walk. Current influenza vaccines protect elderly against viral influenza but not as well as desired. It is expected that the higher doses vaccine can be given with little reaction, but this needs to be tested. Up to 410 people ages 65 years and older will be recruited from the community and from existing volunteer populations. Participants will receive either the high or standard dose injected in the muscle, remain in the clinic for 20 minutes afterward, and maintain a daily memory aid for 7 days. The memory aid will be reviewed by telephone 8-12 days after the injection and return to the clinic or contacted by telephone 6 months after the injection.

DETAILED DESCRIPTION:
Influenza is a common respiratory infection caused by several related viruses. Epidemics of influenza occur each winter and are responsible for an average of about 36,000 deaths each year in the United States. Most of these deaths occur among elderly persons and among people of all ages who suffer from chronic diseases, particularly of the lungs and the heart. Current influenza virus vaccines protect elderly persons against influenza, but not as well as desired. One consideration for trying to increase protection is to increase the vaccine dose, but there is some concern that increasing the dose may increase reactions to the vaccine (such as sore arm, aches, or fever). One of the vaccine manufacturers has prepared an experimental influenza virus vaccine with a dose that is higher than the currently used dose. A previous study with the same high dose of the vaccine showed that it was well tolerated with only increased reactions at the injection site compared to the usual vaccine. Since the study, the high-dose vaccine has also been made without preservative (thimerosal) and gelatin, which are in the standard vaccine. It is expected that this vaccine can be given with little reaction, but this needs to be determined. It also needs to be shown whether such a vaccine stimulates higher levels of infection-fighting proteins (or antibodies) in the blood than standard doses of influenza vaccine. The purpose of this research is to compare reactions and antibody responses following standard flu vaccine to those following the experimental vaccine. Up to 410 people ages 65 years and older will be recruited from the community and from existing volunteer populations. Participants will receive either the high or standard dose injected in the muscle, remain in the clinic for 20 minutes afterward, and maintain a daily memory aid for 7 days. The memory aid will be reviewed by telephone 8-12 days after the injection and return to the clinic or contacted by telephone 6 months after the injection. This study is linked to DMID protocol 05-0028.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for study participation:

* Ambulatory medically stable persons >= 65 years of age on the date of vaccination
* Provides written informed consent and will be available for all study visits
* Able to understand and comply with planned study procedures

Subjects will be considered ambulatory if they are not institutionalized, bedridden, or homebound. Medically stable subjects may have underlying illnesses such as hypertension, diabetes, ischemic heart disease, or hypothyroidism, but their symptoms/signs must be controlled with medical therapy. Subjects with acute febrile illnesses [oral temperature equal to or exceeding 99.5ºF (37.5ºC)] will be deferred until 3 days after illness resolution.

Exclusion Criteria:

Subjects must not meet any of the following exclusion criteria in order to be eligible for participation in this study:

* Known allergy to eggs or other components of the vaccine (eg, thimerosal);
* History of a severe reaction following influenza vaccination, systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing the same substances;
* History of Guillain-Barré Syndrome;
* Immunosuppression as a result of underlying illness or treatment;
* Use of oral steroids, parenteral steroids, or high-dose inhaled steroids (> 800 µg per day of beclomethasone dipropionate or equivalent) within 1 month prior to vaccination;
* Use of other immunosuppressive or cytotoxic drugs or radiation therapy within the six months prior to vaccination;
* Active neoplastic disease or history of any hematologic malignancy in the past 5 years (except localized skin or prostate cancer that is stable in the absence of therapy);
* Acute or chronic condition that (in the opinion of the Investigator) would render vaccination unsafe or would interfere with the evaluation of responses including, but not limited to the following: known chronic liver disease, significant renal disease, oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV, unstable or progressive neurologic disorder, insulin-treated diabetes mellitus;
* Use of experimental vaccines or medications within the month prior to study entry, or expected use of experimental vaccines or medications during the entire study period, including the 6-month follow-up phone call, after inoculation with study vaccine;
* Use of experimental devices or participation in a medical procedure trial within the month prior to study entry, or expected use of experimental devices or participation in a medical procedure trial during the entire study period, including the 6-month follow-up phone call, after inoculation with study vaccine;
* Receipt of immunoglobulin or other blood product within 3 months prior to enrollment;
* Receipt of other licensed vaccines within the preceding 4 weeks or expected to receive a licensed vaccine within 1 month (prior to visit 2) following trial vaccination;
* Subject is enrolled in a conflicting clinical trial;
* Thrombocytopenia or bleeding disorder or therapy contraindicating IM vaccination.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 414 (Actual)
Dates: Start 2005-04; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Iowa - Vaccine Research & Education Unit, Iowa City, Iowa
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Chen WH, Cross AS, Edelman R, Sztein MB, Blackwelder WC, Pasetti MF. Antibody and Th1-type cell-mediated immune responses in elderly and young adults immunized with the standard or a high dose influenza vaccine. Vaccine. 2011 Apr 5;29(16):2865-73. doi: 10.1016/j.vaccine.2011.02.017. Epub 2011 Feb 23. PMID 21352939